CLINICAL TRIAL: NCT04917029
Title: The Efficacy of Adding Dexmedetomidine Perineurally to Bupivacaine in Ultrasound Guided Fascia Iliaca Block Versus Intravenously Infused Dexmedetomidine on Hemodynamic Stability Intraoperatively and Postoperative Analgesia Following Hip Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ismail Mohammed, Lecturer of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: FMASU R 116/2021
Record Dates: First submitted 2021-06-01; First posted 2021-06-08 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active:Group A (Active Comparator): Group A: receive 40 ml bupivacaine 0.25% +5 ml placebo in FICB perineurally in generally anaesthetized patients with intravenous infusion of 0.5 µg/kg/h of Dexmedetomidine.
  Interventions: Drug: Bupivacaine hydrochloride perineurally; Drug: Dexmedetmidine infusion
- (Group B (Active Comparator): Group B: receive FICB with dexmedetomidine 80µg diluted in 5 ml normal saline and 40 ml bupivacaine 0.25% added perineurally in generally anaesthetized patients without dexmedetomidine infusion.
  Interventions: Drug: Bupivacaine hydrochloride perineurally; Drug: Dexmedetomidine perineurally

INTERVENTIONS:
Drug: Bupivacaine hydrochloride perineurally — Arm 1; Bupivacaine hydrochloride 40 ml 0.25% perineurally in FICB
  Other Names: marcaine
Drug: Dexmedetmidine infusion — Arm 1: infusion of Dexmedetmidine 0.5 µg/kg/h
  Other Names: precedex
  Arms: Active:Group A
Drug: Dexmedetomidine perineurally — Arm 2:Dexmedetomidine perineurally in FICB 80µg
  Other Names: precedex
  Arms: (Group B

SUMMARY:
The current study aims to assess effectiveness of dexmedetomidine as adjuvant to general anesthesia on the hemodynamic stability and narcotic consumption intraoperatively and its effect as adjuvant to fascia iliaca compartment block (FICB) with bupivacaine on the postoperative analgesia following hip arthroscopy (decrease the need to narcotics postoperatively avoiding their complications and increasing the success rate of surgery, by enhancing patients to move easier).

DETAILED DESCRIPTION:
This study is a randomized controlled trial at Ain Shams university hospital, Cairo, Egypt. The study will include 88 patients (44 patients) in each group planned for undergoing hip arthroscopy under general anesthesia, will be randomly assigned into one of the following two groups using computer generated codes and opaque sealed envelopes:

All patients will range from ASA I or II, planned for elective hip arthroscopy, aging from 18 to 65 years, body weight renge from 70- 80 Kg of both sexes.

Patients will receive 0.03 mg/kg intravenous (IV) midazolam as a preanesthetic medication, and 1 mg Granisetron as a postoperative nausea and vomiting (PONV) prophylaxis after application of routine monitoring (electrocardiogram, non-invasive blood pressure monitoring and oxygen saturation (SPO2)).

A standard anaesthetic technique will be followed. After preoxygenation for three minutes, anaesthesia will be induced with: propofol 2-3 mg/kg, fentanyl 1µg/kg. Atracuirium besilate 0.5 mg/kg will be used to provide muscle relaxation. All patients will be mechanically ventilated with a tidal volume of 8 ml/kg. 1-2 minimum alveolar concentration (MAC) of isoflurane mixed with oxygen (50%) and air (50%) will be used for maintenance of anesthesia.

GROUP A will receive Dexmedetomidine in dose of of 0.5μg/ kg/hour It elicits a biphasic blood pressure response: a short hypertensive phase followed by hypotension. It is expected that the decreased blood pressure and heart rate, will happen with ongoing therapy within 15 minutes, mediated by central α2A-AR, that decrease the release of noradrenaline from the sympathetic nervous system (10) And that is the reason we will start Dexmedetomidine infusion just after intubation.

Then Ultrasound-guided block was performed in supine position, inguinal ligament was identified, and crease area was sterilized using povidone iodine. Using a 7.5 -12 MHz linear probe, started on the inguinal crease parallel to the inguinal ligament, and after identification of femoral artery, a little movement of the probe laterally till iliopsoas muscle was specified as a hypo echo part in lateral to the artery and femoral nerve. It is covered by a hyperechoic fascia, which separates the muscle from the subcutaneous tissue, using the in-plane technique a 22G/80 mm insulated echogenic block needle was inserted and advanced towards the fascia iliaca and iliopsoas muscle. Confirming the passage of the needle through the fascia iliaca using fascial click and 2mL of saline. LA was injected between fascia iliaca and iliopsoas muscle, we used ultrasound guided hydro dissection technique. Through this hydro dissection, the needle was moved towards the space created by the injected LA. The responsible anesthesiologist and the patient were unaware of the nature of drug in each syringe and master codes were stored by personnel who did not participate in observation.

Mean arterial blood pressure (MABP) and heart rate (HR) will be measured. Any increase or decrease in HR or blood pressure, will be managed as required after exclusion of a surgical cause. For example, MABP or HR rise of > 20% above baseline will be treated by administering a 0.5 μg/kg intravenous bolus of fentanyl.

MABP drop of > 20% below baseline will be dealt with reduction of the isoflurane concentration to 0.6%. If patient is still hypotensive, 6 mg ephedrine will be given intravenously. Finally, bradycardia will be treated with: 0.6 mg IV atropine bolus and repeated as required.

Fentanyl (0.5µg/kg IV) will be titrated intraoperatively at the discretion of the attending anaesthesiologists up to one hour prior to the end of surgery. No other intraoperative adjunct analgesic will be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective hip arthroscopy.
* ASA I and II patients
* aged 18 to 65 years,
* 70-80 kg,
* both sexes.

  * Exclusion Criteria:
* Refusal of the patient to receive FICB or to participate in the study,
* Impaired renal or hepatic functions,
* Asthmatic patients.
* Patients with multiple traumas.
* Obese patients with Body Mass Index > 35.
* Allergy to study drugs.
* Patients with local infection.
* Previous surgery at the injection area.
* Bleeding disorders.
* Patients on anticoagulant therapy,
* Addicts.
* Patients with an opioid analgesic prescription within the last 2 h before the operation.
* Peripheral neuropathy,
* Mental and or psychiatric disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-08-18 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Effect of dexmedetomidine infusion | introperative
  incidence of need rescue agents (fentanyl) intraoperatively and the rate change in heart rate ang blood pressure

SECONDARY OUTCOMES:
Visual Analogue scale (VAS) | 24 hours postoperative
  incidence of need of postoperative analgesic (pethidine) , time of first request and the total dose VAS Will be recorded at 2, 3, 4, 6, 8, 12, 18 and 24 hours. Pethidine 20 mg was administered IV as rescue analgesic if VAS pain score was more than 3 or the patient asked for analgesia and can be repeated after 20 minutes till VAS≤3. The time to first analgesic request and 24 hours total analgesic requirement were recorded and compared. Also, fixed dose of 1 g intravenous acetaminophen will be given /8h.

CONTACTS AND LOCATIONS:
Locations (1):
- Maha Sadek EL Derh, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No